CLINICAL TRIAL: NCT01766557
Title: Assessment of Cod Protein as an Insulin-sensitizing Agent in Women With Polycystic Ovary Syndrome.
Acronym: PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Institute of Nutraceuticals and Functional Foods (Other); Canadian Diabetes Association (Other); Diabetes Québec (Other)
Responsible Party: Principal Investigator, Helene Jacques, Professor, Ph.D., Dt.P., Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PCOS-09-08-078
Record Dates: First submitted 2012-10-02; First posted 2013-01-11 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Insulin Sensitivity; Polycystic Ovarian Syndrome
Keywords: Polycystic ovarian syndrome, sex hormones, ovarian function, women, fish protein, insulin sensitivity, glucose tolerance, β-cell function, inflammation
MeSH Terms: conditions — Insulin Resistance; Polycystic Ovary Syndrome; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semi-controlled intervention with fish protein diet (Experimental): Women with polycystic ovarian syndrome who are assigned to a 12 weeks experimental diet containing cod as the protein source.
  Interventions: Other: Semi-controlled nutritional intervention with fish protein diet
- Semi-controlled intervention with other animal proteins (Active Comparator): Women with polycystic ovarian syndrome who are assigned to a 12 week experimental diet containing beef, pork, veal, eggs and milk products (BPVEM) as protein sources.
  Interventions: Other: Semi-controlled intervention with other animal proteins

INTERVENTIONS:
Other: Semi-controlled nutritional intervention with fish protein diet — After a controlled NCEP-based diet for 3 months, women are assigned to a cod fillet diet. At the end of this first 3 months experimental period, participants return to their NCEP-based diet for a wash-out period of 3 months. Then, each group receive the other diet for an additional 3 months period. The fish protein intake come from cod fillets and correspond to 50% of total protein, the remaining dietary proteins being from BPVEM (20%) and vegetable (30%). Lunches incorporating cod fillets are prepared by professional dietitians, provided two time per week, and are self-consumed. Participants make their breakfasts and dinners using foods from a pre-approved list. Alcohol is strictly prohibited during all periods.
  Arms: Semi-controlled intervention with fish protein diet
Other: Semi-controlled intervention with other animal proteins — Prior to experimental period, participants follow a controlled NCEP-based diet for 3 months. Then women are assigned to a diet containing beef, pork, veal, eggs, milk and milk products. At the end of this first 3 months experimental period, participants return to their NCEP-based diet for a wash-out period of 3 months. The two diets are isoenergetic. The protein intake from BPVEM correspond to 70% of total protein, other dietary proteins are from vegetable (30%) origin. Lunches incorporating animal proteins are prepared by professional dietitians, provided two time per week, and are self-consumed. Participants make their breakfasts and dinners using foods from a pre-approved list. The content in n-3 fatty acids is adjusted to provide equivalent amounts of n-3 fatty acids then in the cod protein diet. Alcohol is strictly prohibited during all periods.
  Arms: Semi-controlled intervention with other animal proteins

SUMMARY:
The objective of our study is to determine the effects of fish protein on insulin sensitivity in PCOS women with insulin resistance, and its mechanism of action on glucose and endocrine metabolism. Our working hypothesis is that dietary fish protein improves insulin sensitivity, glucose tolerance, and related plasma endocrine and lipid abnormalities in PCOS women by restoring secretory β-cell function and insulin signaling to the PI 3-kinase activity/Akt pathway. We further hypothesize that fish protein will improve cycle regularity and ovarian function.

DETAILED DESCRIPTION:
Women with polycystic ovary syndrome are at high risk of developing diabetes. Apart from a primary ovarian defect, up to 10% and 40-50% of those women develop diabetes and insulin resistance (IR) respectively. IR and associated hyperinsulinemia are recognized as important pathogenic factors in determining diabetes in the majority of PCOS women, particularly when obesity is present. Treating IR might reduce the risk of diabetes and improve ovulation and fertility in PCOS women. We recently found that obese, IR men and women consuming a cod protein diet showed a 30% improvement in insulin sensitivity compared with other animal proteins, and also a 24% decrease in high-sensitive C-reactive protein plasma concentration. Therefore, dietary fish protein could represent a natural, safe and practical means to improve insulin sensitivity in PCOS women with IR, and a new non-pharmaceutical approach for the treatment of the multiple endocrine and metabolic abnormalities of PCOS women (see outcome measures for a more extensive description).

ELIGIBILITY:
Inclusion Criteria:

* women
* 18 to 45 years old
* having polycystic ovarian syndrome
* overweight (BMI>27)
* insulin resistance based on fasting insulin levels in the upper 95th percentile (>90pmol/L)
* non-diabetic

Exclusion Criteria:

* diabetes
* hysterectomy
* abnormal endometrial biopsy if abnormal bleeding in the last 6 months
* clinical evidence of Cushing's syndrome
* congenital adrenal hyperplasia (17-OH progesterone>10nmol/l)
* excessive androgens suspicious of a tumour
* prolactins levels >50μg/l
* previous breast, uterus, ovary or liver neoplasia
* use of medication known to affect glucose and lipid metabolisms (e.g. steroid hormones, oral contraceptives, ß-blockers, glitazones, statins, insulin)
* depo-medroxyprogesterone acetate injection in the last year
* important weight loss or weight gain within the last 6 months
* chronic, metabolic (except well controlled chronic hypothyroidism) or acute disease or major surgery within the last 3 months
* dietary incompatibility with calcium supplementation and/or fish consumption (allergy, intolerance, dislike)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in sex hormones, during intervention and from baseline to the end of each intervention period. | At baseline, after the wash-out period, at the end of each intervention period (12 weeks), and at weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11 during the intervention.
  Detailed plasma androgen profile including active androgens (testosterone and dihydrotestosterone), adrenal androgens (androstenedione, dehydroepiandrosterone and its sulphate), major glucuronide-conjugated androgen metabolites, plasma levels of the sex hormone transport protein Sex Hormone-Binding Globulin (SHBG).
Change in cycle regularity during intervention period. | At weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 during the intervention
  menstrual diaries
Change in ovarian function during intervention period. | At weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 during the intervention
  progesterone measurements

SECONDARY OUTCOMES:
Change in nutritional variables from baseline to the end of each intervention period. | At baseline and at the end of the intervention period (12 weeks).
  Food frequency questionnaire
Change in cardiometabolic statute from baseline to the end of each intervention period | At baseline (at the beginning of the intervention), after the 12 weeks wash-out period, and at the end of each intervention period (12 weeks each)
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, glucose and insulin concentrations during a 180-min euglycemic-hyperinsulinemic clamp, GDR, MI, β-cell function, systolic and diastolic blood pressure, glucose and insulin concentrations during a 120-min oral glucose tolerance test, plasma C-peptide concentration, apolipoprotein apoA-1, A-2 and B plasma concentrations, hsCRP, MCP-1, IL-1β, IL-6 and adiponectin concentrations.
Muscle insulin signaling | After each intervention period (12 weeks)
  Muscle biopsies for expression and phosphorylation of IRS-1-associated PI3-K activity, as well as Akt and aPKC activation by insulin.
Change in physical activity habits from baseline to the end of each intervention period. | At baseline and at the end of the intervention period (12 weeks)
  Physical activity habits questionnaire
Change in anthropometric measurements from baseline to the end of each intervention period. | At baseline and at the end of the intervention period (12 weeks)
  anthropometric measurements (body mass index, waist and hip circumferences)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Of Nutraceuticals and Functional Foods (INAF), Laval University, Québec, Quebec, Canada